CLINICAL TRIAL: NCT04290962
Title: African American Cancer Survivor Health: Pilot Implementation Research (National Witness Project® Witness Role Models Use Precision Nutrition)
Brief Title: Web-Based Lifestyle Intervention for the Improvement of Health in African American Cancer Survivors
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no accrual
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: I 77418; NCI-2019-06115 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 77418 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2020-02-27; First posted 2020-03-02 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Cancer Survivor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Supportive Care (web-based lifestyle intervention) (Experimental): Participants complete the 12-month Precision Nutrition Coaching Program web-based lifestyle intervention consisting of physical activity at home or a local gym, nutritional/lifestyle habit with a new focus biweekly, and educational lessons about health, nutrition, fitness, or behavior change.
  Interventions: Behavioral: Lifestyle Therapy; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Behavioral: Lifestyle Therapy — Complete web-based lifestyle intervention
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This early phase I trial studies how well a web-based lifestyle intervention called Precision Nutrition Coaching Program works in improving health in African American cancer survivors. Participating in the web-based lifestyle intervention program reinforced with experienced lifestyle coaches and consisting of physical activity, nutritional/lifestyle habits, and educational lessons may help to improve overall health and well-being, fitness level, and quality of life in African American cancer survivors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To conduct a pilot implementation research study to determine the viability, safety, and effectiveness of the use of a 12-month, commercially available, web-based lifestyle behavioral medicine intervention program by individuals who are or have been a Witness Role Model (WRM) in the National Witness Project (NWP).

SECONDARY OBJECTIVE:

I. To examine the feasibility of this research to subsequently investigate the effects of optimal health and/or lifestyle related behavioral medicine interventions used to promote optimal health on mitigating cancer-related and overall mortality disparities in African Americans (AA), and comorbidity/ chronic disease(s) management over time. (EXPLORATORY)

OUTLINE:

Participants complete the 12-month Precision Nutrition Coaching Program web-based lifestyle intervention consisting of physical activity at home or a local gym, nutritional/lifestyle habit with a new focus biweekly, and educational lessons about health, nutrition, fitness, or behavior change.

ELIGIBILITY:
Inclusion Criteria:

* Has contacted study investigators using the contact information found on recruitment materials to convey their interest in participating
* Verbally confirmed that they now currently or in the past have functioned as a WRM for NWP
* Body mass index (BMI) >= 23
* Weight stable over the past year (=< 10% change)
* Current levels of physical activity were assessed and compared to United States (US) Centers for Disease Control and Prevention (CDC) Physical Activity (PA) guidelines (150 minutes of moderately intensive weekly physical activity)
* Cleared to participate in an exercise program via the American College of Sports Medicine Exercise Pre-participation Health Screening Guidelines
* Has access to internet and a computer/tablet etc
* Has access to basic fitness equipment (dumbbells, resistance bands) and/or is willing to join a fitness facility
* Is currently under the care of and has been assessed by a primary care physician within the last 12 months
* Understands the investigational nature of this study and completes the process of informed consent per Institutional Review Board (IRB) approved protocol

Exclusion Criteria:

* Has uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Is pregnant or nursing
* Is unwilling or unable to participate
* Has any condition which in the investigators' opinion(s) deems the subject an unsuitable candidate to participate in this study
* Has metastatic cancer
* Has an orthopedic disorder, neuromuscular disorder or other condition (e.g., arthritis, morbid obesity) that may significantly preclude participation in exercise or related behaviors
* Is currently incarcerated (i.e., prisoner)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-01-17 (Actual); Primary Completion 2020-10-14 (Actual); Study Completion 2020-10-14 (Actual)

PRIMARY OUTCOMES:
Rate of enrollment | Up to 12 months
Rate of refusal | Up to 12 months
Program adherence rate | Up to 12 months
  Measured by participation and online tracking of activity completion (workout, habit, and lessons). An overall adherence score will be calculated by averaging the percentage of time each of the 3 activities were completed by each participant over the 12-month intervention.
Program retention | Up to 12 months
  Will be measured by the proportion of participants who are still participating in the study at the end of the 12-month intervention.
Incidence of physical activity related injuries | Up to 12 months
  Biweekly inquiries about possible injuries will be conducted.
Program effectiveness | Up to 12 months
  The effects of the lifestyle intervention program will be ascertained via primarily subjective, self-reported assessments administered at pre-intervention, post-intervention, and a follow-up. Subjective data will be validated through the collection of objective data in a subset of local participants via in-person assessments. Generalized linear mixed model methods, specifically a repeated measures analysis of variance with a random participant effect, as well as fixed effects for time and interaction will be used.

OTHER OUTCOMES:
Self-reported cancer related-outcome collection | Up to 12 months
  On line assessments will be completed

CONTACTS AND LOCATIONS:
Overall Officials: Julia Devonish, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States